CLINICAL TRIAL: NCT02176694
Title: Adolescent Controlled Text Messaging to Improve Asthma Medication Adherence in Primary Care.
Acronym: ACT Me
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2013-1184; 1R21HL119826-01 (NIH)
Record Dates: First submitted 2014-06-09; First posted 2014-06-27 (Estimated); Last update posted 2016-06-10 (Estimated); Status verified 2016-06

CONDITIONS: Persistent Asthma
Keywords: persistent asthma; adherence; text message reminders

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Care (No Intervention): Aside from the asthma education provided at enrollment and placement of the SmartInhaler (i.e.,electronic monitoring device), adolescents will continue to receive usual care through their primary care providers.
- Text Messaging (Experimental): A technology based system which allows adolescents to compose, schedule and send one-time or recurring text messages to their own cell phones.
  Interventions: Behavioral: Text Messaging

INTERVENTIONS:
Behavioral: Text Messaging — Website that allows adolescents to create, schedule and send one-time or recurring text messages that will serve as a reminder to take asthma medication or follow up with another health-related matter.
  Arms: Text Messaging

SUMMARY:
A randomized controlled trial of a texting intervention to increase adherence to preventative asthma medication in four Cincinnati Children's Hospital Medical Center primary care clinics.

DETAILED DESCRIPTION:
Our first aim is to determine the feasibility, acceptability and use of a low intensity text messaging intervention to improve adherence to inhaled corticosteroid (ICS) therapy among high risk adolescents with persistent asthma. Our second aim is to determine effect sizes of the intervention to improve adherence (As measured by electronic monitoring and self-report); clinical asthma control; and asthma related quality of life among adolescents with persistent asthma. Our third and final aim is to determine the temporal relationship between text message receipt and ICS canister actuation in order to understand mechanisms by which text messaging may increase ICS adherence.

ELIGIBILITY:
Inclusion Criteria:

* provider-diagnosed persistent asthma
* prescription of an ICS in accordance in NHLBI Expert Panel Report 3 guidelines for at least 30 days prior to enrollment
* Asthma Control Test (ACT) score less than 20 (indicating lack of current control)
* no provider-diagnosed exacerbation in the 30 days prior to enrollment
* possession of a text-enabled cell phone and a plan to keep it throughout the study period
* agreement by parents (or participants over 18 years old) to any charges levied by their cell phone carrier for text messages associated with the study if they do not have an unlimited texting plan
* speak and read English

Exclusion Criteria:

* another chronic lung disease (which would complicate measurement of asthma control)
* cognitive or psychiatric disorder that the treating clinician judges would impair study participation
* use of Advair diskus for their ICS (for which no reliable electronic monitor exists)
* current enrollment in another asthma intervention study

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 29 (Actual)
Dates: Start 2014-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Objective Adherence to ICS | Baseline
  Electronic monitor logs
Change in objective adherence to ICS | Change from baseline in objective adherence to ICS at 1 month
  Electronic Monitor Logs
Change in objective adherence to ICS | Continuous change over time from baseline in objective adherence to ICS at 2 months in intervention compared to control
  Electronic Monitor Logs
Change in objective adherence to ICS | Continuous change over time from baseline in objective adherence to ICS at 3 months in intervention compared to control
  Electronic Monitor Logs
Change in objective adherence to ICS | Continuous change over time from baseline in objective adherence to ICS at 4 months in intervention compared to control
  Electronic Monitor Logs
Change in objective adherence to ICS | Continuous change over time from baseline in objective adherence to ICS at 5 months in intervention compared to control
  Electronic Monitor Logs
Feasibility, Acceptability and Usability of the Text Messaging Website | At time of text messaging intervention
  The Computer System Usability Questionnaire is a self-reported measure that captures quantitative data about the usability of the computer system. The Cincinnati Bell Usability questionnaire is a self-reported measure that captures quantitative and qualitative data about how easy the system is to use, whether they like using it, as well as likes and dislikes. Use of the computer system is determined through CMSText website login and message logs.
Feasibility, Acceptability and Usability of the Text Messaging Website | up to 1 month after receiving text messages
  The Computer System Usability Questionnaire is a self-reported measure that captures quantitative data about the usability of the computer system. The Cincinnati Bell Usability questionnaire is a self-reported measure that captures quantitative and qualitative data about how easy the system is to use, whether they like using it, as well as likes and dislikes. Use of the computer system is determined through CMSText website login and message logs.
Feasibility, Acceptability and Usability of the Text Messaging Website | up to 2 months after receiving text messages
  The Computer System Usability Questionnaire is a self-reported measure that captures quantitative data about the usability of the computer system. The Cincinnati Bell Usability questionnaire is a self-reported measure that captures quantitative and qualitative data about how easy the system is to use, whether they like using it, as well as likes and dislikes. Use of the computer system is determined through CMSText website login and message logs.
Feasibility, Acceptability and Usability of the Text Messaging Website | up to 3 months after receiving text messages
  The Computer System Usability Questionnaire is a self-reported measure that captures quantitative data about the usability of the computer system. The Cincinnati Bell Usability questionnaire is a self-reported measure that captures quantitative and qualitative data about how easy the system is to use, whether they like using it, as well as likes and dislikes. Use of the computer system is determined through CMSText website login and message logs.

SECONDARY OUTCOMES:
Asthma Control | Baseline
  The Asthma Control Test (ACT) are questions that ask about frequency of day and night symptoms, frequency of fast acting inhaler use, environmental triggers, limitations of activities, perception of asthma control, and confidence in ability to manage asthma.
Change in Asthma Control | Change from Baseline at 1 month
  The Asthma Control Test (ACT) are questions that ask about frequency of day and night symptoms, frequency of fast acting inhaler use, environmental triggers, limitations of activities, perception of asthma control, and confidence in ability to manage asthma.
Change in Asthma Control | Continuous change over time from baseline at 2 months in intervention compared to control
  The Asthma Control Test (ACT) are questions that ask about frequency of day and night symptoms, frequency of fast acting inhaler use, environmental triggers, limitations of activities, perception of asthma control, and confidence in ability to manage asthma.
Change in Asthma Control | Continuous change over time from baseline at 3 months in intervention compared to control
  The Asthma Control Test (ACT) are questions that ask about frequency of day and night symptoms, frequency of fast acting inhaler use, environmental triggers, limitations of activities, perception of asthma control, and confidence in ability to manage asthma.
Change in Asthma Control | Continuous change over time from baseline at 4 months in intervention compared to control
  The Asthma Control Test (ACT) are questions that ask about frequency of day and night symptoms, frequency of fast acting inhaler use, environmental triggers, limitations of activities, perception of asthma control, and confidence in ability to manage asthma.
Change in Asthma Control | Continuous change over time from baseline at 5 months in intervention compared to control
  The Asthma Control Test (ACT) are questions that ask about frequency of day and night symptoms, frequency of fast acting inhaler use, environmental triggers, limitations of activities, perception of asthma control, and confidence in ability to manage asthma.
Asthma Symptoms, Quality of Life, Treatment Barriers | Baseline
  The Pediatric Quality of Life (PEDSQL) Asthma Symptom Scale, the generic core scale and the treatment barriers scale are questions that assess how much asthma has been a problem for them in the last month.
Change in Asthma Symptoms, Quality of Life, Treatment Barriers | Change from Baseline at month 1
  The Pediatric Quality of Life (PEDSQL) Asthma Symptom Scale, the generic core scale and the treatment barriers scale are questions that assess how much asthma has been a problem for them in the last month.
Change in Asthma Symptoms, Quality of Life, Treatment Barriers | Continuous change over time from baseline at 2 months in intervention compared to control
  The Pediatric Quality of Life (PEDSQL) Asthma Symptom Scale, the generic core scale and the treatment barriers scale are questions that assess how much asthma has been a problem for them in the last month.
Change in Asthma Symptoms, Quality of Life, Treatment Barriers | Continuous change over time from baseline at 3 months in intervention compared to control
  The Pediatric Quality of Life (PEDSQL) Asthma Symptom Scale, the generic core scale and the treatment barriers scale are questions that assess how much asthma has been a problem for them in the last month.
Change in Asthma Symptoms, Quality of Life, Treatment Barriers | Continuous change over time from baseline at 4 months in intervention compared to control
  The Pediatric Quality of Life (PEDSQL) Asthma Symptom Scale, the generic core scale and the treatment barriers scale are questions that assess how much asthma has been a problem for them in the last month.
Change in Asthma Symptoms, Quality of Life, Treatment Barriers | Continuous change over time from baseline at 5 months in intervention compared to control
  The Pediatric Quality of Life (PEDSQL) Asthma Symptom Scale, the generic core scale and the treatment barriers scale are questions that assess how much asthma has been a problem for them in the last month.

CONTACTS AND LOCATIONS:
Overall Officials: Maria T. Britto, M.D., M.P.H., Principal Investigator — Professor of Pediatrics
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] Dodds CM, Britto MT. Learnings from a pragmatic pilot trial of text messaging for high-risk adolescents with asthma. Ann Allergy Asthma Immunol. 2018 May;120(5):546-547. doi: 10.1016/j.anai.2018.02.008. Epub 2018 Feb 9. No abstract available. PMID 29432968